CLINICAL TRIAL: NCT02365948
Title: A Randomized, Double-blind, Placebo-controlled, Single Escalating Dose Study of Subcutaneous Certolizumab Pegol (CZP) to Evaluate the Pharmacokinetics and Safety of CZP in Healthy Chinese Subjects
Brief Title: A Study of Certolizumab Pegol to Evaluate Pharmacokinetics and Safety in Adult Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA0045
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Certolizumab Pegol; Healthy Chinese subjects
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Certolizumab Pegol 100 mg (Experimental): Subjects will receive100 mg of CZP given by subcutaneous injections in healthy Chinese subjects. The dose group begins treatment on Day 1.
  To achieve an injectable CZP 100 mg dose, a manual process will be applied by the unblinded site pharmacist.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- Certolizumab Pegol 200 mg (Experimental): Subjects will receive 200 mg of CZP given by subcutaneous injections in healthy Chinese subjects. The dose group begins treatment staggered by a minimum of 14 days from CZP 100 mg. Dose escalation will be suspended according to the predefined criteria and process.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- Certolizumab Pegol 400 mg (Experimental): Subjects will receive 400 mg of CZP (two injections of CZP 200 mg) given by subcutaneous injections in healthy Chinese subjects. The dose group begins treatment staggered by a minimum of 14 days from CZP 200 mg. Dose escalation will be suspended according to the predefined criteria and process.
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- Placebo (Placebo Comparator): For assessment of the Adverse Event (AE) profile, there are 2 placebo controls in each dose group. The placebo subjects receive the injection of saline (NaCl 0.9 %) at the same time (and of the same volume) as the CZP subjects.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active Substance: Certolizumab Pegol
  * Pharmaceutical Form: Prefilled syringes
  * Concentration: 200 mg/mL
  * Route of Administration: Subcutaneous injection
  Other Names: Cimzia; CDP870; CZP
  Arms: Certolizumab Pegol 100 mg; Certolizumab Pegol 200 mg; Certolizumab Pegol 400 mg
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Prefilled syringes
  * Concentration: 0.9 % Saline
  * Route of Administration: Subcutaneous injection
  Other Names: PBO

SUMMARY:
This study will characterize the pharmacokinetics (PK) of certolizumab pegol (CZP) and evaluate safety of CZP in healthy Chinese subjects. 36 subjects will be randomized to receive one of 3 dose levels of CZP or placebo. The total study duration will be approximately 71-94 days for each subject.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-center, single escalating dose study in healthy Chinese subjects. The primary objective of the study is to characterize the pharmacokinetics (PK) of certolizumab pegol (CZP) in healthy Chinese subjects after a single subcutaneous (sc) dose. The secondary objective is to evaluate safety of CZP in healthy Chinese subjects after a single sc dose. 36 healthy Chinese subjects (18 male and 18 female) will be randomized to receive one of 3 dose levels of CZP (100 mg, 200 mg and 400 mg) or placebo given by sc injections. Each dose group begins treatment staggered by a minimum of 14 days. The total duration of the study will be approximately 71 to 94 days for each subject. This includes a 2 to 21 days Screening Period, 1 day of treatment and 70 days Observation Period after administration of a single dose of investigational medicinal product.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) / Independent Ethics Committee (IEC) approved written Informed Consent Form (ICF) is signed and dated by the subject
* Subject is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule or medication intake according to the judgment of the investigator
* Subject is male or female between 18 and 45 years of age, inclusive
* Results of clinical laboratory tests within the reference range of the laboratory or outside the reference range of the laboratory but considered as nonclinically significant by the investigator. This is not allowed for aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) and bilirubin values above the upper limit of normal (ULN) ranges
* Have a body weight of 50 to 80 kg and a body mass index (BMI) between 19 and 24 kg/m^2
* In good health as determined by the investigator on the basis of medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) and results of laboratory tests during the Pretreatment Period (Screening and Baseline)
* Nonsmoker and former smoker who have given up smoking more than 6 months before first administration
* Willing to abstain from alcohol-, tobacco- and caffeine-containing products for 48 hours prior to admission into the clinic and during the entire in-clinic stay
* Subjects should be a registered permanent Citizen of the People's Republic of China and are Chinese as evidenced by all 4 grandparents as Chinese by ethnical definition
* Female subjects of childbearing potential should have negative pregnancy test at Screening and at Baseline (Day -1) and should use a medically accepted method of contraception (one barrier method and including another - ie, hormonal contraception for at least 2 cycles, intrauterine device, implant device, diaphragm with spermicide, monogamous relationship with vasectomized [for at least 3 months] partner or using condoms with spermicide gel) during the entire duration of the study

Exclusion Criteria:

* Active malignancies or a history of malignancy, excluding basal cell carcinoma of the skin that had been excised prior to study start
* History of adverse reaction to polyethylene glycol
* History of severe or multiple allergies
* Known Tuberculosis (TB) disease, high risk of acquiring TB infection, or latent TB infection
* A history of chronic infection, recent serious or life-threatening infection (within 6 months, including herpes zoster), or a current sign or symptom that may indicated an infection
* Subject with a history or active systemic / respiratory infection due to fungal, parasitic, or mycotic pathogens including but not limited to histoplasmosis, coccidiosis, paracoccidiosis, pneumocystis, blastomyces, aspergillus, and nontuberculous mycobacteria
* History of an infected joint prosthesis at any time with prosthesis still in situ
* Positive hepatitis B surface antigen, hepatitis C Virus immunoglobulin G (HCV IgG), or Human Immunodeficiency Virus (HIV) test result during the Screening
* Subject with blood pressure and pulse rate (measured in supine position, after 10 minutes rest) outside the normal range
* A mean corrected QT interval using Bazett's formula (QTcB) interval >450 ms at Screening. If the mean QTcB exceeds the limits above, one additional triplicate electrocardiogram (ECG) may be taken. If this triplicate also gives an abnormal result, the subject should be excluded
* Any history or evidence of any clinically significant (CS) cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy, or any other CS abnormality, as judged by the investigator
* History of substance abuse, drug addiction or alcoholism within 3 years prior to Screening
* Inability to abstain from smoking during the in-clinic stay
* Subject has made a blood donation or had a comparable blood loss (>350 mL) within the last 3 months prior to first intake of study drug
* Positive result of alcohol test or urine drug Screen
* Receiving any other Investigational Medicinal Product (IMP) within 3 months or 5 half-lives of it, whichever is longer, prior to the first dose of IMP or is scheduled to receive an IMP other than CZP during the course of the study
* Previous exposure to or has participated in studies with any other anti-TNFα antibody (Ab) compounds
* Use of any medication, prescription or over-the-counter within 14 days or 5 half-lives of the medication, whichever is longer, before the first dose of IMP, or it is anticipated to need any medication during the study
* Has been on herb medication during the last 2 weeks prior to screening, or is currently taking it
* Excessive use of caffeine-containing beverages exceeding 500 mg caffeine/day (5 cups of coffee)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve from time zero up to the last analytically quantifiable concentration (AUC 0-t) | D1 (pre-dose and 1, 2, 4, 8, 12 hrs post-dose), D2 (24, 36 hrs post-dose), D3 (48 hrs post-dose), D4 (72 hrs post-dose), D5 (96 hrs post-dose), D6, D8, D15, D22, D29, D43, D57 and D70
  AUC 0-t is within a period of 70 days following the dose of CZP, reported in units of μg/mL·h, as determined using the linear trapezoidal rule.
Maximum plasma concentration (Cmax) | D1 (pre-dose and 1, 2, 4, 8, 12 hrs post-dose), D2 (24, 36 hrs post-dose), D3 (48 hrs post-dose), D4 (72 hrs post-dose), D5 (96 hrs post-dose), D6, D8, D15, D22, D29, D43, D57 and D70
  The maximum observed plasma concentration of CZP.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero up to infinity (AUC) | D1 (pre-dose and 1, 2, 4, 8, 12 hrs post-dose), D2 (24, 36 hrs post-dose), D3 (48 hrs post-dose), D4 (72 hrs post-dose), D5 (96 hrs post-dose), D6, D8, D15, D22, D29, D43, D57 and D70
  AUC is calculated as AUC=AUC(0-t)+Clast/λz, where Clast is the last quantifiable plasma concentration and λz is the apparent terminal elimination rate constant.
Time to reach a maximum plasma concentration (Tmax) | D1 (pre-dose and 1, 2, 4, 8, 12 hrs post-dose), D2 (24, 36 hrs post-dose), D3 (48 hrs post-dose), D4 (72 hrs post-dose), D5 (96 hrs post-dose), D6, D8, D15, D22, D29, D43, D57 and D70
  The time of occurrence of Cmax.
Terminal half-life (t½) | D1 (pre-dose and 1, 2, 4, 8, 12 hrs post-dose), D2 (24, 36 hrs post-dose), D3 (48 hrs post-dose), D4 (72 hrs post-dose), D5 (96 hrs post-dose), D6, D8, D15, D22, D29, D43, D57 and D70
  t½ is reported in units of hours, as determined via simple linear regression (slope=-λz) of natural log(ln) concentration vs time for data points in the terminal phase of the concentration-tim curve. t½ is calculated as ln(2)/λz.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 1, Shanghai, China